CLINICAL TRIAL: NCT02217280
Title: Dispersal Pattern of Injectate After Cervical Epidural Steroid Evaluated With Magnetic Resonance Imaging
Brief Title: Dispersal Pattern for Spine Injections (Gadolinium Contrast)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Christina Goldstein, Principal Investigator, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1210810
Record Dates: First submitted 2014-03-21; First posted 2014-08-15 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Gadolinium; gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection with Gadolinium (Experimental): This group of patients identified by the PI as having cervical radiculopathy will receive gadolinium (the intervention) in their epidural cervical injection along with steroid (DepoMedrol). There is no control group in this study.
  Interventions: Drug: Injection with Gadolinium

INTERVENTIONS:
Drug: Injection with Gadolinium — Gadavist (gadobutrol) injection is a gadolinium-based contrast agent indicated for intravenous use in diagnostic magnetic resonance imaging (MRI) in adults and children (2 years of age and older) to detect and visualize areas with disrupted blood brain barrier (BBB) and/or abnormal vascularity of the central nervous system
  Other Names: Gadavist

SUMMARY:
This study will analyze injectate dispersal patterns after standard-of-care cervical epidural steroid injections using gadolinium as a marker and magnetic resonance imaging (MRI) to characterize the pattern. Although these procedures are performed with high frequency under the assumption that injectate remains localized to injection site, no peer-reviewed studies have validated this assumption. Comprehensive characterization of injectate dispersal patterns will provide important data regarding safety, as well as diagnostic and therapeutic potential of cervical epidural steroid injections.

DETAILED DESCRIPTION:
Epidural steroid injections have long had an impact in the treatment of various spine-related conditions, particularly radiculopathy. The efficacy of epidural spinal injections has been attributed to the anatomic location reached by the injectate. Cervical epidural steroid injections are also used as an injury location indicator. This application is based on documenting pain relief after injection into a specific location in the cervical spine. Both the diagnostic and therapeutic applications for epidurals assume that the injectate remains local to the injection site in order to have its effects. However, in a recently completed study, the investigators group documented substantial diffusion of injectate after lumbar epidurals used computerized tomography (CT) assessments.1 Based on the exposure to ionizing radiation associated with CT along with the superior imaging specificity and sensitivity of MRI, the investigators are shifting their imaging modality to MRI for future studies. The proposed study is designed to evaluate the use of gadolinium and MRI to assess nature and amount of diffusion of injectate in the cervical region after standard-of-care epidural injections. To the investigators knowledge, this will be the first study to critically assess this common procedure in order to evaluate safety and efficacy in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Cervical radiculopathy patient as identified by principle investigator

Exclusion Criteria:

* Patients unable to give consent or comply with rehabilitation process
* Pregnant
* Co-morbidities such as infection, malignancy, myelopathy or an uncontrolled medical condition
* Allergy to injectate
* Anticoagulative state
* Severe claustrophobia
* Non-MRI compatible pacemaker, neurostimulator, bladder stimulator or other mechanical device
* Renal disease that would cause the patient to be at an increased risk of complication of receiving the contrast agent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Goldstein, MD, Principal Investigator — University of Missouri Department of Orthopaedics
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical ESI With Gadolinium: Male and female subjects between the ages of 18-85 with cervical radiculopathy as identified by the study PI. This was a single arm study with a one-time cervical interlaminar injection at the C7-T1 level. A total injection dose of 10.1 ml included 0.1 mL of gadolinium, 2 ml of 10 mg/ml dexamethasone and 8 ml normal saline, which was administered under fluoroscopic guidance.
Period: Overall Study
Arm/Group | Cervical ESI With Gadolinium
Started | 20
Completed | 16
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Post-consent sceen fail | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cervical ESI With Gadolinium
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 51.18 [39 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Injection Dispersal Patterns Measured (in cm) in the Superoinferior Directions on Post-injection MRI With a Calibrated Internal Measurement Software.
Description: Determine the relative efficacy (diagnostic and therapeutic) of cervical epidural injections based on injectate diffusion. We will measure (with post-injection MRI) how far the injection travels in the superoinferior directions (in cm) within in the epidural space.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Injection With Gadolinium
Number analyzed (Participants) | 16
cm | 14.73 (3.15)

2. Primary Outcome: Circumferential Contrast Spread
Description: Number of study subjects who achieved circumferential contrast spread in the epidural space. Circumferential contrast spread is achieved when the contrast reaches all directions in the epidural space in the horizontal/axial plane.
  This includes contrast spread in the anterior, posterior, medial and lateral directions (in relation to the spinal cord).
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Groups:
- Cervical ESI: Male and female subjects between the ages of 18-85 with cervical radiculopathy. This was a single arm study.
Arm/Group | Cervical ESI
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: 1 year
Description: Regular investigator assessment
Arm/Group | Cervical ESI With Gadolinium
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No